CLINICAL TRIAL: NCT05700292
Title: Effect of High-intensity Interval Training on Low-grade Systemic Inflammation in Obese Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-60
Record Dates: First submitted 2022-05-03; First posted 2023-01-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: High-intensity Interval Training; Systemic Inflammation; Obesity
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Training (Experimental): Training is based on 5 circuits, with intervals of 1 minute (high intensity) by 2 minutes (low intensity), with a total training time of 15 minutes (plus 5 more minutes of warm-up and 5 of cool-down exercises). The high intervals will be performed with the following exercises: squat, reverse lunge & knee-up, reverse jump and walkout pushup, while the low intervals were performed jogging. The heart rates of the study subjects will be calculated using the Astrand test and the progression criteria is going to be based on an increase in maximum heart rate of 85% to 95%. To monitor heart rate during training, a polar brand chest sensor, model H9, will be used.
  Interventions: Other: High-intensity Interval Training
- Moderate-intensity continuous training (Active Comparator): Continuous aerobic training (jogging). Also, the heart rates of the study subjects will be calculated using the Astrand test and the progression criteria is going to be based on an increase in maximum heart rate from 60% to 75% and an increase in training time from 25 to 45 minutes (considering 5 minutes of warm-up and 5 of cool-down exercises). To monitor heart rate during training, a polar brand chest sensor, model H9, will be used as well.
  Interventions: Other: Moderate-intensity continuous training

INTERVENTIONS:
Other: High-intensity Interval Training — Training is based on 5 circuits, with intervals of 1 minute (high intensity) by 2 minutes (low intensity), with a total training time of 15 minutes (plus 5 more minutes of warm-up and 5 of cool-down exercises). The high intervals will be performed with the following exercises: squat, reverse lunge & knee-up, reverse jump and walkout pushup, while the low intervals were performed jogging. The heart rates of the study subjects will be calculated using the Astrand test and the progression criteria is going to be based on an increase in maximum heart rate of 85% to 95%. To monitor heart rate during training, a polar brand chest sensor, model H9, will be used.
  Arms: High-intensity Interval Training
Other: Moderate-intensity continuous training — Continuous aerobic training (jogging). Also, the heart rates of the study subjects will be calculated using the Astrand test and the progression criteria is going to be based on an increase in maximum heart rate from 60% to 75% and an increase in training time from 25 to 45 minutes (considering 5 minutes of warm-up and 5 of cool-down exercises). To monitor heart rate during training, a polar brand chest sensor, model H9, will be used as well.
  Arms: Moderate-intensity continuous training

SUMMARY:
Background: Obesity is a multifactorial disease that affects 36% of the Mexican population; it is characterized by the excessive accumulation of adipose tissue in the body, mainly in the abdominal region, conditions that are closely linked to low-grade systemic inflammation (LGSI). Scientific evidence suggests that LGSI can be attenuated by the benefits of regular physical exercise, since such activity has the potential to decrease the concentrations of certain proinflammatory molecules, such as reactive C protein, tumor necrosis factor alpha and interleukin 6. Objective: To analyze the LGSI response when intervening with a high-intensity interval training in young obese adults between 18 to 30 years. Materials and methods: The present study is defined as a simple randomized clinical trial. Participants will be randomized into one of two groups of intervention; 1: High-intensity interval training (HIIT), and the control group with moderate-intensity continuous training (MICT). The interventions will be 3 times a week for 2 months, completing a total of 24 sessions. The HIIT group will carry out the activities at high intensity (85 to 95% maximum heart rate) aerobic type training; density of 1 minute at high interval followed by 2 minutes of low interval with a total time of 15 minutes (plus 5 more minutes of warm-up and 5 of cool-down exercises). While the MICT group will carry out the activities with a moderate intensity (60 to 75% maximum heart rate) aerobic type training reaching a total time of 25 to 45 minutes (considering 5 minutes of warm-up and 5 of cool-down exercises). Physical activity will be monitored using a Polar brand heart rate sensor (model H9). Anthropometric, biochemical, and inflammatory assessments will be monitored at baseline, at 4 weeks (mid-intervention), and at 8 weeks (end of intervention). Biochemical parameters will be determined by dry chemistry (Vitros 350), anthropometry by electrical bioimpedance (Inbody 370), and inflammatory markers by blood count and ProQuantum Immunoassay technology. Infrastructure: Institute of Translational Nutrigenomics and Nutrigenomics, University Center for Health Sciences, University of Guadalajara.

DETAILED DESCRIPTION:
Detailed description Hypothesis High-intensity interval training decreases inflammatory markers associated with low-grade chronic systemic inflammation in obese young adults aged 18 to 30 years.

Methods Study design Simple randomized clinical trial. Location of the study. Institute of Translational Nutrigenomics and Nutrigenomics of the Department of Molecular Biology and Genomics of the University Center for Health Sciences and at the Tlajomulco University Center of the University of Guadalajara.

Virtual environment: ZOOM

Sample size:

The sample size was determined according to the mean difference formula for clinical trials from a previous study (Barrón et. al, 2020), with a confidence percentage of 95%, statistical power of 90% and alpha of 5%. The sampling is extended to a potentially larger amount of 20% to avoid the negative impact of the results due to the dropout rate of the study subjects. The sample required for each group results from a minimum of 13 subjects per group. Therefore, an "n" of 16 patients per group will be captured.

Group 1: HIIT Group 2 (control): MICT Study subjects An invitation will be made to participate in this project by facebook, whatsapp, Instagram, tiktok and physical posters which will be placed in the Civil Hospital of Guadalajara "Fray Antonio Alcalde" and in the University Science Center of Guadalajara. Health (CUCS). Subjects who decide to accept must go to the Institute of Translational Nutrigenomics and Nutrigenomics, they will undergo a clinical and anthropometric assessment, and if they meet the inclusion criteria, their authorization will be requested through their signature on an informed consent letter.

Clinical evaluation A medical checkup will aim to assess the general health status of the participant by a qualified professional to identify possible health risks. The biomechanical evaluation will look for alterations related to the musculoskeletal system that prevent the practice of certain motor gestures of the participant. The biomechanical evaluation will be carried out by a qualified Physiotherapist with a title and professional license. A submaximal stress test based on the Astrand-Ryhming protocol (Astrand, 1954) will be performed on a cycle ergometer with electronic brake (RECK MOTOmed) to determine the maximum oxygen consumption and maximum heart rate with the aim of structuring the individualized physical activity program. Anthropometric measurements (weight, height, waist circumference, hip circumference) will be made by a certified Anthropometrist with reference to the ISAK protocol (The International Society for the Advancement of Kinanthropometry). The percentages of body fat and muscle mass will be obtained by the electrical bioimpedance method with the Inbody 370.

Biochemical analysis Participants who pass the previous filter will proceed to the baseline evaluation, which will be carried out 7 days prior to the start of the intervention.

For the evaluation of the blood count and cytokines in plasma, fasting for 8 to 12 hours will be requested; venous puncture of the antecubital region will be performed with a 21 French caliber catheter. Samples will be collected in dry or EDTA vacutainer tubes (BD Vacutainer) to be centrifuged for 10 min at 4°C at 3500 rpm. TNFalpha and IL-6 will be analyzed using the ProQuantum Immunoassay technique based on the instructions proposed by the manufacturer.

Randomization The assignment of the study groups will be defined using the simple random method. The first subject who meets the inclusion criteria will be selected as a starting point to be included in group A, then the second subject will be assigned to group B, and so on until the total "n" of the study is reached. Subjects with odd numbers (1, 3, 5…) will be assigned to group A, and subjects with even numbers (2, 4, 6…) will be assigned to group B.

Biochemical determinations Blood samples will be obtained in the morning after an 8 to 10 hour fast. Total cholesterol (TC), HDL cholesterol and triglycerides (TG) values will be determined using a VITROS® 350 dry chemistry kit (Ortho Clinical Diagnostics, Buckinghamshire, England); the LDL-c value will be calculated using the Friedewald formula, the TG/HDL ratio will be obtained by dividing the TG values by the HDL-c values.

Anthropometric evaluation Height will be evaluated with a SECA portable stadiometer (Hamburg, Germany) with a precision of 1 mm and a precision of 0.5 cm. Subjects will be positioned with their head oriented in the Frankfort plane, with their heels, buttocks and back in contact with the scale and feet together. Waist circumference will be obtained using a Lufkin (USA) tape measure following the guidelines of the International Society for the Advancement of Kinanthropometry (ISAK). The cut-off point that will be used for its interpretation will be that reported by the NCEP/ATPIII (<88cm in women and <102cm in men). The percentage of body fat (PBF) interpretation will be: adequate <25% in men and <35% in women.

Intervention The beginning and development of the intervention will be developed in a virtual environment through "ZOOM". Indications will be given through a brochure with recommendations for a balanced diet, based on the current recommendations of the WHO (World Health Organization, 2018). Participants from both groups will be trained and conditioned for 2 weeks prior to the start of training.

The interventions will be for 12 weeks, 3 times a week completing 24 total sessions. The appointment schedule for the initial evaluation, which will be held at the University Center for Health Sciences of the University of Guadalajara, taking into account the conditions of the pandemic and strengthening the security measures in terms of health risks. It should be noted that the training will be monitored by specialists in Physical Activity and Rehabilitation Sciences.

The HIIT model is built from a series of free isotonic aerobic exercises adapted to the characteristics of the participants and based on the recommendations of the guidelines for the performance and monitoring of high-intensity interval training in clinical populations (Taylor et al. ., 2019) and a previous trial (Gallo-Villegas el al, 2018).

Reassessment A first assessment will be made in relation to the clinical, anthropometric and biochemical evaluation at week 6 (half of the intervention) and the final at week 12. The post tests will be carried out 72 hours after the last training session to avoid biases associated with acute exercise response. The procedures will be faithfully reproduced.

Determination of TNFalpha, IL-6 and reactive C protein concentrations The serum concentrations of TNFα, IL-6 will be determined by means of the ProQuantum Immunoassay technique, for the determinations of cytokines such as: TNFalpha (A35601), IL-6 (A35573), the ProQuantum Immunoassay methodology will be used, which starts from the antigen antibody binding methodology, in this case the antibody will be coupled to oligonucleotide chains that, when bound to the antigen, will be close enough for a ligase to join them and generate a template DNA base and thereby begin the PCR amplification process real time, in the Light Cycler 96 equipment. The serum concentration of ultrasensitive reactive C protein will be determined by means of an immunoassay with the getein equipment.

Databases and computer programs The sociodemographic data, the values of the anthropometric variables and the biochemical variables will be captured in the Microsoft Excel 2010 program for later statistical analysis in the IBM SPSS software (Statistical Package for the Social Sciences, Chicago IL.) for Windows version 21.

Statistical analysis For the normality distribution of the variables, the Kolmogorov-Smirnov test will be used. For the descriptive analysis, the qualitative variables will be expressed as frequency and percentage and the quantitative variables as mean and standard deviation. For the comparative analysis of the parametric quantitative variables between two groups, a Student's t test will be performed and an ANOVA test between three groups, followed by an analysis with post-hoc tests. Regarding the evaluation of the individual and joint effect of two or more risk factors on a quantitative dependent variable, the linear regression model will be used. A confidence interval of 95% will be considered and a value of p<0.05 will be considered as statistically significant in each of the tests.

Biosecurity considerations For the planning and development of this research, the standards of Good Clinical Practices (GCP) have been considered, which were presented in 1994 by the International Conference on Harmonization, which provide a guarantee for the study subjects that their rights, safety and well-being are protected at all times.

Related to biosafety, it is going to be followed the statements of official Mexican standards NOM-087-ECOL-SSA1-2002 for issues related to the management and disposal of infectious biological material, and NOM-052-SEMARNAT-2005 for the management and disposal of material identified in hazardous waste.

Ethical considerations In accordance with the Regulation of the General Law of Health in the Matter of Research for Health 1987, in the second title, on the ethical aspects of research in human beings, chapter 1, article 17, the protocol is classified as research with risk minimum.

The determinations of the Official Mexican Standard NOM-004-SSA3-2012 of the clinical file will be considered, which establishes that the data of the participants must be confidential. Each participant will be given the corresponding informed consent, which will explain in detail the characteristics of the study, its objectives, the methodology for collecting information, benefits and consequences of their participation, as well as the confidentiality and dissociation of the data. data that you provide us and that obtained through the analysis of the blood sample; the latter in accordance with articles 18, 19 and 21 of the Federal Law of Transparency and Access to Public and Government Information. Additionally, the use of the General Law on Protection of Personal Data Held by Obliged Entities is supported, as well as the Declaration of Helsinki.

The benefits for the participants will be feedback on their body composition and general recommendations for healthy lifestyle.

The information obtained will be used for research and will only be accessed by the research team. The identification data of the participants will not appear in the publications derived from the project, to maintain and guarantee their anonymity and confidentiality.

Moreover, the main researcher and the collaborators of this study do not declare any conflicts of interest that influence the results, recruitment, retention of participants, publication of data and ethical review of the project.

This study has been already accepted by the ethics committee of the Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, with the CI-06321 number.

ELIGIBILITY:
Inclusion Criteria:

* Young adults, between 18 and 30 years.
* BMI ≥ 30-39.9 kg/m2
* How signed the informed consent
* Additionally, it is necessary that they have computer equipment, electronic tablet, or smart cell phone, as well as access to electricity and the Internet.

Exclusion Criteria:

* Participants who smoke
* Presence of any of the following comorbidities: hypothyroidism, type 1 diabetes mellitus, type 2 diabetes mellitus, arterial hypertension, oncological pathology, immunological or rheumatic diseases.
* Consumption of nitrates and anticalcium drugs during the 4 days prior to the start of the investigation and beta blockers, hypoglycemic drugs 7 days prior to the start of the intervention.
* Pregnant or breastfeeding
* Men who consume more than 40 g/day of alcohol or women who consume more than 20 g/day
* Postural and biomechanical alterations (knee, foot or spine)
* Previous diagnosis and less than 6 months of COVID 19
* Previous diagnosis of HIV +
* Previous diagnosis of periodontal disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum levels of IL-6 between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity. | Change from baseline of IL-6 at 4 and 8 weeks
  Compare serum levels of IL-6 between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity.

SECONDARY OUTCOMES:
Waist circumference between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years. | Change from baseline of waist circumference between a high-intensity interval training vs moderate-intensity continuous training at 4 and 8 weeks
  Compare the waist circumference (cm) between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years.
Serum levels of TNFα between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity. | Change from baseline of TNFα at 4 and 8 weeks
  Compare serum levels of TNFα between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity.
Serum levels of ultrasensitive reactive C protein between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity. | Change from baseline of ultrasensitive reactive C protein at 4 and 8 weeks
  Compare serum levels of ultrasensitive reactive C protein between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity.
Serum levels of erythrocyte sedimentation rate between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity. | Change from baseline of erythrocyte sedimentation rate at 4 and 8 weeks
  Compare serum levels of erythrocyte sedimentation rate between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity.
Serum levels of neutrophil-lymphocyte ratio between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity. | Change from baseline of neutrophil-lymphocyte ratio at 4 and 8 weeks
  Compare serum levels of neutrophil-lymphocyte ratio between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity.
Waist-hip ratio between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years. | Waist-hip ratio between a high-intensity interval training vs moderate-intensity continuous training at 4 and 8 weeks
  Waist-hip ratio (waist (cm)/ hip (cm)) between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years.
BMI between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years. | BMI between a high-intensity interval training vs moderate-intensity continuous training at 4 and 8 weeks
  BMI (kg/m2) between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years.
Body fat between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years. | Body fat and muscle mass percentage between a high-intensity interval training vs moderate-intensity continuous training at 4 and 8 weeks
  Body fat between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years.
Muscle mass percentage between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years. | Muscle mass percentage between a high-intensity interval training vs moderate-intensity continuous training at 4 and 8 weeks
  Muscle mass percentage between a high-intensity interval training vs moderate-intensity continuous training in young adults with obesity between 18 and 30 years.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Martinez-Lopez, PhD, Principal Investigator — University of Guadalajara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abd El-Kader SM, Al-Jiffri OH. Aerobic exercise modulates cytokine profile and sleep quality in elderly. Afr Health Sci. 2019 Jun;19(2):2198-2207. doi: 10.4314/ahs.v19i2.45. PMID 31656505
- [Background] Ahn N, Kim K. Can Active Aerobic Exercise Reduce the Risk of Cardiovascular Disease in Prehypertensive Elderly Women by Improving HDL Cholesterol and Inflammatory Markers? Int J Environ Res Public Health. 2020 Aug 14;17(16):5910. doi: 10.3390/ijerph17165910. PMID 32824020
- [Background] ASTRAND PO, RYHMING I. A nomogram for calculation of aerobic capacity (physical fitness) from pulse rate during sub-maximal work. J Appl Physiol. 1954 Sep;7(2):218-21. doi: 10.1152/jappl.1954.7.2.218. No abstract available. PMID 13211501
- [Background] Barron-Cabrera E, Gonzalez-Becerra K, Rosales-Chavez G, Mora-Jimenez A, Hernandez-Canaveral I, Martinez-Lopez E. Low-grade chronic inflammation is attenuated by exercise training in obese adults through down-regulation of ASC gene in peripheral blood: a pilot study. Genes Nutr. 2020 Aug 27;15(1):15. doi: 10.1186/s12263-020-00674-0. PMID 32854610
- [Background] Feito Y, Heinrich KM, Butcher SJ, Poston WSC. High-Intensity Functional Training (HIFT): Definition and Research Implications for Improved Fitness. Sports (Basel). 2018 Aug 7;6(3):76. doi: 10.3390/sports6030076. PMID 30087252
- [Background] Gallo-Villegas J, Aristizabal JC, Estrada M, Valbuena LH, Narvaez-Sanchez R, Osorio J, Aguirre-Acevedo DC, Calderon JC. Efficacy of high-intensity, low-volume interval training compared to continuous aerobic training on insulin resistance, skeletal muscle structure and function in adults with metabolic syndrome: study protocol for a randomized controlled clinical trial (Intraining-MET). Trials. 2018 Feb 27;19(1):144. doi: 10.1186/s13063-018-2541-7. PMID 29482601
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Fisher G, Brown AW, Bohan Brown MM, Alcorn A, Noles C, Winwood L, Resuehr H, George B, Jeansonne MM, Allison DB. High Intensity Interval- vs Moderate Intensity- Training for Improving Cardiometabolic Health in Overweight or Obese Males: A Randomized Controlled Trial. PLoS One. 2015 Oct 21;10(10):e0138853. doi: 10.1371/journal.pone.0138853. eCollection 2015. PMID 26489022
- [Background] Furuncuoglu Y, Tulgar S, Dogan AN, Cakar S, Tulgar YK, Cakiroglu B. How obesity affects the neutrophil/lymphocyte and platelet/lymphocyte ratio, systemic immune-inflammatory index and platelet indices: a retrospective study. Eur Rev Med Pharmacol Sci. 2016 Apr;20(7):1300-6. PMID 27097950
- [Background] Ihalainen JK, Schumann M, Eklund D, Hamalainen M, Moilanen E, Paulsen G, Hakkinen K, Mero AA. Combined aerobic and resistance training decreases inflammation markers in healthy men. Scand J Med Sci Sports. 2018 Jan;28(1):40-47. doi: 10.1111/sms.12906. Epub 2017 Jun 13. PMID 28453868